CLINICAL TRIAL: NCT05268133
Title: Aronia and Cognitive Fitness: Focus on Brain Insulin-Sensitivity and Vascular Function
Brief Title: Aronia and Cognitive Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 21-084
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-10

CONDITIONS: Brain Vascular Function; Cognition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aronia (Experimental): An aronia melanocarpa extract. Study volunteers will receive a daily oral dose of 160 mg AME for 6 weeks.
  Interventions: Dietary Supplement: Aronia
- Control (Placebo Comparator): Cellulose. Study volunteers will receive a daily oral dose of 160 mg cellulose for 6 weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Aronia — As described in experimental arm
  Arms: Aronia
Dietary Supplement: Control — As described in placebo comparator arm
  Arms: Control

SUMMARY:
Previously, beneficial effects of Aronia Melanocarpa extract (AME) supplementation on cognitive performance has been observed in healthy middle-aged adults. However, underlying mechanisms have not yet been addressed. In addition, effects of AME are unknown in subjects at increased risk of cognitive impairment. It is hypothesized that supplementation with AME enhances (regional) brain vascular function and brain insulin-sensitivity, thereby improving cognitive function of subjects at increased risk of cognitive impairment.

The primary objectives are to investigate effects of AME intake on brain vascular function and insulin-sensitivity in cognitive-control brain areas, while we will also evaluate changes in cognitive function (secondary objective).

The present study is a randomized, double-blind, placebo-controlled, cross-over trial consisting of two study groups and a pre- and post-test day in both study arms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 55-75 years
* BMI between 25-35 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Smoking or smoking cessation < 12 months
* Presence of diabetes mellitus
* Active cardiovascular disease like congestive heart failure or cardiovascular event
* Severe medical conditions, including asthma, chronic obstructive pulmonary disease (COPD), kidney failure, auto-inflammatory diseases or rheumatoid arthritis
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use of dietary supplements or medication affecting the main outcomes of the study
* Use of an investigational product within another biomedical intervention trial within the previous month
* Contra-indications for MRI imaging (e.g., pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)
* Left-handedness
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use medication to treat blood pressure, lipid or glucose metabolism

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Brain Vascular function | Change after 6 weeks of intervention
  cerebral blood flow as quantified non-invasively by the MRI perfusion method arterial spin labeling (ASL MRI). Higher cerebral blood flow indicates improved brain vascular function.
Brain insulin sensitivity | Change after 6 weeks of intervention
  cerebral blood flow as quantified non-invasively by the MRI perfusion method arterial spin labeling (ASL MRI) before and after application of intranasal insulin (160 IU).
  Higher cerebral blood flow after intranasal insulin application indicates improved brain insulin sensitivity

SECONDARY OUTCOMES:
Cognitive performance | Change after 6 weeks of intervention
  Quantified through the Cambridge Neuropsychological Test Automated Battery (CANTAB).

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University
Locations (1):
- Metabolic Research Unit Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahles S, Plat J, Nijssen KM, Joris PJ. Aronia melanocarpa extract supplementation affects brain vascular function and cognitive performance: A randomized, double-blind, placebo-controlled, cross-over study in older adults with overweight or obesity. Clin Nutr. 2026 Feb;57:106561. doi: 10.1016/j.clnu.2025.106561. Epub 2025 Dec 29. PMID 41499921